CLINICAL TRIAL: NCT00973856
Title: Evaluation of the Effectiveness of an Alcohol Based Hand Gel for the Reduction of Warts on the Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Clinic Akron General (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09025
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Papillomavirus Infections; Warts; Condylomata Acuminata; Epidermodysplasia Verruciformis
MeSH Terms: conditions — Papillomavirus Infections; Warts; Condylomata Acuminata; Epidermodysplasia Verruciformis | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- PURELL Left Hand/ Placebo Right Hand (Experimental): One product will be assigned to each hand to minimize treatment confusion for the participants.
  PURELL VF481 Left Hand/ Placebo Right Hand
  Interventions: Other: PURELL VF481; Other: Placebo Solution
- Placebo Solution Left Hand/ PURELL Right hand (Placebo Comparator): One (1) product will be assigned to each hand to minimize treatment confusion for the participants PURELL VF481 Right Hand/ Placebo Left Hand
  One (1) pump of test product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
  Interventions: Other: PURELL VF481; Other: Placebo Solution

INTERVENTIONS:
Other: PURELL VF481 — One (1) pump of test product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
  Other Names: PURELL VF481 alcohol based hand gel
Other: Placebo Solution — One (1) pump of product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed

SUMMARY:
The objective is to conduct a pilot study to determine the effectiveness of PURELL VF481 to treat warts located on the hands.

DETAILED DESCRIPTION:
* At least 5, but not more than 20 participants will be enrolled in the study.
* Each wart is randomly assigned a test product prior to the start of the study
* Warts are equally distributed between products so that an equal number of warts treated on each person. One (1) product will be assigned to each hand to minimize treatment confusion for the participants
* The test product will be applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage.
* Subjects will log date and time of application and anything notable (such as changes in wart appearance or missed dose) in a log book.
* Measurement of wart (longest diameter) and photos taken at each visit by trained office medical assistants, LPNs, PA-C or MD.
* Time points for office visitation: Baseline (0 weeks), 4 weeks, 8 weeks, 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients with 2+ warts being seen at a Dermatologist's office
* 2 or more warts on the hands that are located at least 1 cm apart or on separate fingers
* Warts must have been present for at least 2 months
* Wart size must be between 2 mm-15 mm in diameter
* Participants must be in good general health
* Participants must be able to speak and read in English.
* Participant must be able to read and sign participant instruction sheet, and informed consent and authorization.
* Subjects must be able to understand and execute the instructions presented in pictorial form.

Exclusion Criteria:

* Pregnancy (Patients will be asked to verify using criteria of contraception, menstrual cycle, and pregnancy test, if necessary).
* Treatment of warts with other methods such as salicylic acid, etc., in the past 14 days.
* Known allergies to common topical antimicrobials or the individual ingredients in either test product.
* Participation in a clinical study in the past 7 days or participation in another clinical study
* Unwillingness to perform requirements of the study
* Any medical condition that should preclude participation in the study, at the discretion of the physician
* Missed ≥ 6 of the treatments in a 4 week study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliot Mostow, M.D>, Principal Investigator — Cleveland Clinic Akron General
Locations (1):
- Akron Dermatology, Akron, Ohio, United States

REFERENCES:
- See also: Akron General Medical Center — http://www.akrongeneral.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no pre-assignment details. Once consented, pts were enrolled into both study arms.
Units Other Than Participants: warts,not pts assigned to intervention
Groups:
- PURELL VF481 Left Hand/ Placebo Right Hand: Warts are equally distributed between products so that an equal number of warts treated on each person. One (1) product will be assigned to each hand to minimize treatment confusion for the participants
  PURELL VF481: One (1) pump of test product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
- Placebo Solution Left Hand/ PURELL VF481 Right Hand: Warts are equally distributed between products so that an equal number of warts treated on each person One (1) product will be assigned to each hand to minimize treatment confusion for the participants
  One (1) pump of test product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
  Placebo Comparator: One (1) pump of product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
Period: Overall Study
Arm/Group | PURELL VF481 Left Hand/ Placebo Right Hand | Placebo Solution Left Hand/ PURELL VF481 Right Hand
Started | 3; 5 warts,not pts assigned to intervention | 2; 5 warts,not pts assigned to intervention
Completed | 3; 5 warts,not pts assigned to intervention | 2; 5 warts,not pts assigned to intervention
Not Completed | 0; 0 warts,not pts assigned to intervention | 0; 0 warts,not pts assigned to intervention

BASELINE CHARACTERISTICS:
Units Other Than Participants: warts
Groups:
- Placebo Solution Left Hand/ PURELL VF481 Right Hand: Warts are equally distributed between products so that an equal number of warts treated on each person. One (1) product will be assigned to each hand to minimize treatment confusion for the participants
  One (1) pump of test product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
  Placebo Comparator: One (1) pump of product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
- Total: Total of all reporting groups
Arm/Group | PURELL VF481 Left Hand/ Placebo Right Hand | Placebo Solution Left Hand/ PURELL VF481 Right Hand | Total
Number analyzed (Participants) | 3 | 2 | 5
Number analyzed (warts) | 5 | 5 | 10
Age, Categorical [Count of Units; unit: warts]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Units; unit: warts]
  Sex/Gender unspecified | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Difference in % Reduction in Wart Size Between Product A and Product B at Each Timepoint
Description: Data is not available due to study closure and data destruction
Time Frame: Baseline, 4, 8, and 12 weeks, change at 12 weeks reported
Population: Data is not available due to study closure and data destruction
Units Other Than Participants: wart reduction %
Groups:
- Purell VF481: Active Ingredient: 70% ethanol
Arm/Group | Purell VF481
Number analyzed (Participants) | 0
Number analyzed (wart reduction %) | 0

2. Secondary Outcome: Change in Size of Warts Treated by Each Product at Each Time Point.
Description: Data is not available due to study closure and data destruction
Time Frame: Baseline, 4, 8 and 12 weeks, change at 12 weeks reported
Population: Data is not available due to study closure and data destruction
Groups:
- PURELL Left Hand/ Placebo Right Hand: One product will be assigned to each hand to minimize treatment confusion for the participants.
  PURELL VF481 Left Hand/ Placebo Right Hand
  PURELL VF481: One (1) pump of test product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
  Placebo Solution: One (1) pump of product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
- Placebo Solution Left Hand/ PURELL Right Hand: One (1) product will be assigned to each hand to minimize treatment confusion for the participants PURELL VF481 Right Hand/ Placebo Left Hand
  One (1) pump of test product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
  PURELL VF481: One (1) pump of test product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
  Placebo Solution: One (1) pump of product (approximately 1.5ml) is applied to a wooden applicator and gently rubbed into the wart, then covered with a latex free adhesive bandage (it is not necessary to wait until dry) each night before bed
Arm/Group | PURELL Left Hand/ Placebo Right Hand | Placebo Solution Left Hand/ PURELL Right Hand
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Same definition
Groups:
- Placebo: 15% alcohol formulation that aesthetically resembles VF481
Arm/Group | Purell VF481 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No